CLINICAL TRIAL: NCT04314440
Title: Cognitive Processing in Preterm Infants and NICU Music Therapy
Acronym: NICU-MT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Saskatchewan Health Authority - Regina Area (Other)
Collaborators: University of Regina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: REB15-100
Record Dates: First submitted 2016-03-17; First posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Other Preterm Infants
Keywords: Cognitive; Preterm; Infants; Music; Therapy; NICU
MeSH Terms: conditions — Premature Birth | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Music therapy (Experimental): After the initial warm up session music therapy will be delivered three times a week for 15-20 minutes. All babies in the experimental group will be exposed to three weeks of music therapy sessions that is a total of 9 music therapy session prior to discharge from the hospital. The baby will be placed at the bassinet 15 minutes before music therapy begins. The baby will be in the bassinet during music therapy and 15 minutes post music therapy to allow measurement of physiological indicators. If parents are present during music therapy they will not engage in kangaroo care during the music therapy session or when physiological measurements are being taken pre and post music therapy, but can do so at other times.
  Interventions: Behavioral: Music therapy
- Control (No Intervention): Infants in this group will not receive any music therapy but will receive all other standard care provided to infants at the Regina General Hospital (RGH). All measurements will be carried out for all the infants in this group at the time when observations are carried out for infants in the music therapy group.

INTERVENTIONS:
Behavioral: Music therapy — An accredited music therapist will deliver 15-20 minutes of music therapy every day, 4-5 days in week one and remaining in week two to all MT participants. All participants in music therapy group will get a total of nine sessions. The lullaby "twinkle twinkle little star" will be sung for ~5 minutes, followed by the same songs played on acoustic guitar for ~5 minutes and another ~5 minutes of the same song sung in voice. This protocol will be followed in all 9 sessions for all infants in the experimental arm. The sound levels will be maintained at 55-65 decibels (dB) using appropriate meters. If MT is interrupted within 10 minutes then a make-up session will be delivered, assuming no discharge. In case of missed sessions and interrupted session infants will receive a maximum of 12 session.
  Arms: Music therapy

SUMMARY:
Several positive physiological and behavioural outcomes have been observed in preterm infants exposed to music therapy during their stay at Neonatal Intensive Care Units (NICU). There is ample evidence in the literature showing that brief exposure to music can lead to superior performance on a host of cognitive tasks in laboratory settings in children, adolescent and adults. However, till date no study has examined the cognitive benefits of NICU music therapy in preterm infants. Further habituation tests have been employed to examine cognitive functioning in infants in laboratory setting but the same test have not been employed as a measure to examine early cognitive functioning in preterm infants.

This project will be carried out to examine the benefits of NICU music therapy on the cognitive functioning of preterm infants born at 27- 33 weeks of gestational age. A randomized controlled research design will be employed to compare cognitive functioning between the treatment and control group at 18 - 24 months of corrected gestational age. The treatment group will be exposed to music therapy during their stay in NICU and the controlled group will be exposed to all standardized care available at our institution except music therapy. Habituation tests will be used to examine cognitive functioning of the preterm infants in groups at 18 - 24 months of gestational age.

DETAILED DESCRIPTION:
Following previous research, our hypothesis is that infants in the experimental group will display significantly more positive scores on a collection of physiological and behavioural measurements. The stimuli used at each age will be targeted to the infants' developmental level. Bayley Scales of Infant Development will also be administered at 18 - 24 months as part of high risk infant follow up. These data will be included in the analysis for outcome measurement. While seated in a high-chair or their parent's lap, infants will be habituated to a series of images of a particular shape (e.g., a triangle), while their looking time to each stimulus is measured. Each image during habituation will be a unique token of the category (i.e., all different triangles). Habituation will be individually determined, and defined as cumulative looking across three successive trials that is 50% than cumulative looking across the first three trials. Following habituation, infants will be shown a novel token of the habituation shape (e.g., a new triangle) and a novel shape (e.g., a square), in counterbalanced order. If infants recognize the category change, they should look longer at novel category compared to the novel token. For each test, two dependent measures will be sampled: rate of habituation and amount of dishabituation to the novel category. Mixed ANOVA and paired t-tests will be used to analyze the data. As preterm infants have been shown to be delayed on these kinds of tasks, we hypothesize that the experimental group will habituate to each category faster, and/or display stronger dishabituation scores compared to the preterm. We will also use multiple regression analyses to examine relations between the NICU physiological and behavioural measures and the cognitive measures. We hypothesize that infants who most strongly benefited from their therapies in the NICU will display the most advanced cognitive abilities. An intention-to-treat- analysis will be performed for cognitive measures as well. The cognitive assessment at 2 and 4 months that were to be carried out at the Developmental Lab at University of Regina is now canceled due to feasibility concerns.

ELIGIBILITY:
Inclusion Criteria:

1. Gestation age 27-33 weeks (maternal dates or early fetal ultrasound)
2. Is not on ventilators
3. Written informed consent forms has been signed from the infant's legal guardian

Exclusion Criteria:

1. Infants with congenital abnormalities
2. Severe intraventricular hemorrhage, with ventriculomegaly or parenchymal hemorrhage
3. Infants with known or suspected prenatal exposure to substance
4. Infants receiving palliative care at NICU
5. Infants who are on ventilators
6. Infants whose legal guardian did not sign the consent forms

Ages: 27 Weeks to 33 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 102 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Time looking at a familiar stimulus | 18 - 24 months
  Average difference in rate of habituation as measure by the time looking at a familiar stimulus in mili-seconds between experimental and control groups.

SECONDARY OUTCOMES:
Physiological measure | 15 minutes,before, during, after music therapy, 6 days a week
  Average difference in heart rate before music therapy to after music therapy from before to during and from during to after music therapy.
Physiological measure | 15 minutes,before, during, after music therapy, 6 days a week
  Average difference in breathing rate before music therapy to after music therapy from before to during and from during to after music therapy.
Physiological measure | 15 minutes,before, during, after music therapy, 6 days a week
  Average difference in oxygen saturation before music therapy to after music therapy from before to during and from during to after music therapy.
Behavioral measure | Before to after music therapy 6 days a week
  Difference in sleep between experimental and control group
Behavioral measure | Before to after music therapy 6 days a week
  Difference in apnea between experimental and control group
Behavioral measure | Before to after music therapy 6 days a week
  Difference in Bradycardia (number and severity) between experimental and control group
Behavioral measure | Before to after music therapy 6 days a week
  Difference in de-saturation degree of it between experimental and control group

OTHER OUTCOMES:
Other outcomes | Baseline to 3 weeks when music therapy is complete
  Average difference in weight gain (total calorie intake) between experimental and control group
Other outcome | Baseline
  Average difference in length of hospitalization between experimental group and control group
Other outcome | Baseline
  Average difference in neurological assessment score between experimental group and control group
Other outcome | Baseline
  Average difference in hearing assessment between experimental group and control group

CONTACTS AND LOCATIONS:
Overall Officials: Jayalakshmi Bodani, Principal Investigator — Saskatchewan Health Authority - Regina Area
Locations (1):
- Regina General Hospital, Neonatal Intensive Care Unit, Deaprtment of Pediatrics, Regina, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: Yes